CLINICAL TRIAL: NCT01667562
Title: Phase IIIb, Open-Label Study of Erlotinib (Tarceva®) Treatment in Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer Who Present Activating Mutations in the Tyrosine Kinase Domain of the Epidermal Growth Factor Receptor
Brief Title: A Study of Erlotinib in Participants With Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Acronym: ESSENCE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML27860
Record Dates: First submitted 2012-08-15; First posted 2012-08-17 (Estimated); Results first posted 2019-12-20 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride

ARMS (2):
- Erlotinib (Experimental): Erlotinib will be administered as a single daily oral dose of 150 milligrams until disease progression, death or unacceptable toxicity.
  Interventions: Drug: Erlotinib
- Diagnostic Phase (No Intervention): Participants with advanced or metastatic NSCLC were tested for EGFR mutations. Participants who did not have an EGFR mutation were excluded from the study.

INTERVENTIONS:
Drug: Erlotinib — Daily oral doses administered until disease progression or unacceptable toxicity or death.
  Other Names: Tarceva
  Arms: Erlotinib

SUMMARY:
This open-label, multi-center study will evaluate the progression-free survival and safety of erlotinib in participants with locally advanced or metastatic non-small cell lung cancer with activating mutations in the tyrosine kinase domain of the epidermal growth factor receptor (EGFR). Participants will receive daily oral doses of erlotinib until disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of locally advanced or metastatic non-small cell lung cancer with activating mutations in the tyrosine kinase domain of the EGFR
* Measurable disease according to RECIST
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Life expectancy greater than or equal to (>/=) 12 weeks
* Adequate hematological, liver and renal function
* Participants with asymptomatic and stable cerebral metastases receiving medical treatment

Exclusion Criteria:

* Previous chemotherapy or treatment against EGFR for metastatic disease
* Treatment with an investigational agent less than 3 weeks before enrollment
* History of neoplasm other than non-small cell lung cancer (except carcinoma in situ of the uterine cervix, basal cell skin carcinoma, or prostate carcinoma)
* Participants with symptomatic cerebral metastases
* Any significant ophthalmologic abnormality
* Unstable systemic disease
* Coumarins use
* Evidence of any other disease, neurological or metabolic dysfunction, physical examination or laboratory finding contraindicating the use of an investigational drug
* Participants with pre-existing parenchymal lung disease such as pulmonary fibrosis, lymphangiosis carcinomatosis
* Participants with known infection with human immunodeficiency virus (HIV), Hepatitis B (HBV), Hepatitis C (HCV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2012-01-20 (Actual); Primary Completion 2017-09-07 (Actual); Study Completion 2017-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- Serbia (4):
  - Clinic for Pulmonology, Clinical Center of Serbia, Belgrade
  - Clinical Center Bezanijska Kosa; Oncology, Belgrade
  - Institute for pulmonary diseases of Vojvodina, Kamenitz
  - Clinical Center Nis; Clinic for pulmonary diseases Knez Selo, Niš

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 375 participants were in the diagnostic population. Out of the 375 participants, only 30 participants had EGFR mutation and were eligible for erlotinib treatment.
Groups:
- Erlotinib: Erlotinib was administered as a single daily oral dose of 150 milligrams until disease progression, death or unacceptable toxicity.
Period: Diagnostic Phase
Arm/Group | Diagnostic Phase | Erlotinib
Started | 375 | 0
Completed | 345 | 0
Not Completed | 30 | 0
Not completed — Started Erlotinib in Treatment Period | 30 | 0
Period: Erlotinib Phase
Arm/Group | Diagnostic Phase | Erlotinib
Started | 0 | 30
Completed | 0 | 27
Not Completed | 0 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Switch to Commercial Drug | 0 | 1

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population included all participants enrolled in the study.
Groups:
- Baseline Population: Participants with advanced or metastatic NSCLC were tested for EGFR mutations and enrolled in the study.
Arm/Group | Baseline Population
Number analyzed (Participants) | 375
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 375 participants were in the diagnostic population. Out of the 375 participants, only 30 participants had EGFR mutation and were eligible for erlotinib treatment.
  years
    Diagnostic Phase | 62.2 (9.2)
    Erlotinib: number analyzed (Participants) | 30
    Erlotinib | 62.4 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 375 participants were in the diagnostic population. Out of the 375 participants, only 30 participants had EGFR mutation and were eligible for erlotinib treatment.
  Participants
    Diagnostic Phase: Female | 133
    Diagnostic Phase: Male | 242
    Erlotinib: number analyzed (Participants) | 30
    Erlotinib: Female | 18
    Erlotinib: Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 375 participants were in the diagnostic population. Out of the 375 participants, only 30 participants had EGFR mutation and were eligible for erlotinib treatment.
  Participants
    Diagnostic Phase: American Indian or Alaska Native | 0
    Diagnostic Phase: Asian | 0
    Diagnostic Phase: Native Hawaiian or Other Pacific Islander | 0
    Diagnostic Phase: Black or African American | 0
    Diagnostic Phase: White | 375
    Diagnostic Phase: More than one race | 0
    Diagnostic Phase: Unknown or Not Reported | 0
    Erlotinib: number analyzed (Participants) | 30
    Erlotinib: American Indian or Alaska Native | 0
    Erlotinib: Asian | 0
    Erlotinib: Native Hawaiian or Other Pacific Islander | 0
    Erlotinib: Black or African American | 0
    Erlotinib: White | 30
    Erlotinib: More than one race | 0
    Erlotinib: Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival as Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 (v 1.1)
Description: Kaplan Meier estimate of the median PFS was defined as the time at which half of the participants have progressed (progressive disease [PD]) based on RECIST tumor response criteria or died from any cause, whichever occurred first. PD: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Patients who had not died or progressed at the time of the final analysis were censored at the date of last contact.
Time Frame: Baseline until disease progression, or death, whichever occurs first (approximately up to 4 years and 9 months)
Population: The intent-to-treat population included all participants enrolled in the study. There were no patients excluded from analysis either in efficacy and safety analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib
Number analyzed (Participants) | 30
months | 9.574 [5.525 to 13.662]

2. Secondary Outcome: Proportion of Participants With Objective Response as Assessed by RECIST v 1.1
Description: Objective response (OR) was based on criteria related to changes in size of target lesions according to modified RECIST. Target lesions were selected on the basis of their size (lesions with the longest diameter) as well as the feasibility of reproducible repeated measurements. OR was the sum of complete response (CR) and partial response (PR) four at least 4 weeks during treatment. CR: disappearance of all target lesions. PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: Baseline until disease progression, or death, whichever occurs first (approximately up to 4 years and 9 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 30
proportion of participants | 0.67 [0.49 to 0.81]

3. Secondary Outcome: Proportion of Participants With Disease Control as Assessed by RECIST v 1.1
Description: Disease control was defined as objective response or stable disease (SD) for at least 6 weeks. OR was based on criteria related to changes in size of target lesions according to modified RECIST. Target lesions were selected on the basis of their size (lesions with the longest diameter) as well as the feasibility of reproducible repeated measurements. OR was the sum of CR and PR four at least 4 weeks during treatment. CR: disappearance of all target lesions. PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: Baseline until disease progression, or death, whichever occurs first (approximately up to 4 years and 9 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 30
proportion of participants | 0.97 [0.82 to 1.00]

4. Secondary Outcome: Proportion of Participants With Epidermal Growth Factor Receptor (EGFR) Mutations
Description: Mutations in the EGFR included exon 19 deletion mutations and the single-point substitution mutation L858R in exon 21.
Time Frame: Screening up to approximately 7 days
Population: This study had 2 phases: 1st phase - included 375 patients assessed for EGFR mutations 30 patients (out of these 375) had EGFR mutations and they were included in 2nd phase - treatment with Erlotinib.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Diagnostic Phase
Number analyzed (Participants) | 375
proportion of participants | 0.08 [0.06 to 0.11]

5. Secondary Outcome: Percentage of Participants With Adverse Events
Description: An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Baseline up to approximately 4 years and 9 months
Population: The safety population was identical to the ITT population, which included all participants enrolled in the study.
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 30
percentage of participants | 76.7

6. Secondary Outcome: Change From Baseline to End of Study in Quality of Life Score Using The Functional Assessment of Cancer Therapy Lung (FACT-L)
Description: The domains in the Quality of life score using the Functional Assessment of Cancer Therapy Lung (FACT-L) include physical, social/family, emotional, and functional well-being, and a lung cancer subscale include symptoms, cognitive function and regret of smoking. Minimum and maximum value of the scale is 0 and 4, respectively. Higher score indicate better health state.
Time Frame: Baseline and end of study (approximately 4 years and 9 months)
Population: Participants without disease progression who filled out the FACT-L questionnaire.
Measure: Mean (Standard Deviation); unit: unit on a scale
Arm/Group | Erlotinib
Number analyzed (Participants) | 1
unit on a scale | -2.83 (NA) — The standard deviation could not be calculated for one participant who had data for this outcome.

ADVERSE EVENTS:
Time Frame: 4 years and 9 months
Description: The safety population was identical to the ITT population. The ITT population comprised all 30 patients.
Arm/Group | Erlotinib
All-Cause Mortality (participants affected / at risk) | 1/30
Serious Adverse Events (participants affected / at risk) | 6/30
Other Adverse Events (participants affected / at risk) | 22/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=30)
Rash (Skin and subcutaneous tissue disorders) | 3
Paronychia (Skin and subcutaneous tissue disorders) | 1
Death (General disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=30)
Rash (Skin and subcutaneous tissue disorders) | 14
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2
Fatigue (General disorders) | 4
Anemia (Blood and lymphatic system disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-08-16): https://cdn.clinicaltrials.gov/large-docs/62/NCT01667562/Prot_SAP_000.pdf